CLINICAL TRIAL: NCT01961921
Title: A Phase 2, Multicenter, Open-Label, Extension Study to Evaluate the Long-Term Safety, Clinical Activity, and Pharmacokinetics of ALN-TTR02 in Patients With Familial Amyloidotic Polyneuropathy Who Have Previously Received ALN-TTR02
Brief Title: The Study of ALN-TTR02 (Patisiran) for the Treatment of Transthyretin (TTR)-Mediated Amyloidosis in Patients Who Have Already Been Treated With ALN-TTR02 (Patisiran)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALN-TTR02-003; 2013-001644-65 (EudraCT Number)
Record Dates: First submitted 2013-10-09; First posted 2013-10-14 (Estimated); Results first posted 2018-10-30 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2018-11

CONDITIONS: TTR-mediated Amyloidosis
Keywords: RNAi therapeutic
MeSH Terms: interventions — patisiran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ALN-TTR02 (patisiran) (Experimental)
  Interventions: Drug: ALN-TTR02 (patisiran) administered by intravenous (IV) infusion

INTERVENTIONS:
Drug: ALN-TTR02 (patisiran) administered by intravenous (IV) infusion

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of long-term dosing with ALN-TTR02 (patisiran) in patients with transthyretin (TTR) mediated amyloidosis (ATTR).

ELIGIBILITY:
Inclusion Criteria:

* Previously received and tolerated ALN-TTR02 (patisiran) in Study ALN-TTR02-002.
* Adequate Karnofsky performance status, liver function, and renal function.

Exclusion Criteria:

* Pregnant or nursing.
* Has had a liver transplant.
* Has a New York Heart Association heart failure classification >2.
* Has unstable angina.
* Has uncontrolled clinically significant cardiac arrhythmia.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-10; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jared Gollob, MD, Study Director — Alnylam Pharmaceuticals
Locations (9):
- Clinical Trial Site, Boston, Massachusetts, United States
- Clinical Trial Site, Rio de Janeiro, Brazil
- France (2):
  - Clinical Trial Site, Le Kremlin-Bicêtre
  - Clinical Trial Site, Marseille
- Clinical Trial Site, Münster, Germany
- Portugal (2):
  - Clinical Trial Site, Lisbon
  - Clinical Trial Site, Porto
- Clinical Trial Site, Palma de Mallorca, Spain
- Clinical Trial Site, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Access to Anonymized individual participant data that support these results is made available 12 months after study completion and not less than 12 months after the product and indication have been approved in the US and/or the EU.
  Data will be provided contingent upon the approval of a research proposal and the execution of a data sharing agreement. Requests for access to data can be submitted via the website www.vivli.org.

REFERENCES:
- [Derived] Coelho T, Adams D, Conceicao I, Waddington-Cruz M, Schmidt HH, Buades J, Campistol J, Berk JL, Polydefkis M, Wang JJ, Chen J, Sweetser MT, Gollob J, Suhr OB. A phase II, open-label, extension study of long-term patisiran treatment in patients with hereditary transthyretin-mediated (hATTR) amyloidosis. Orphanet J Rare Dis. 2020 Jul 8;15(1):179. doi: 10.1186/s13023-020-01399-4. PMID 32641071

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 27 subjects were enrolled.
Groups:
- ALN-TTR02 (Patisiran): Patients received 0.3 mg/kg of ALN-TTR02 (patisiran) every three weeks
Period: Overall Study
Arm/Group | ALN-TTR02 (Patisiran)
Started | 27
Completed | 25
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: All patients who received at least one dose of ALN-TTR02 (patisiran)
Arm/Group | ALN-TTR02 (Patisiran)
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (15.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 18
Familial Amyloidotic Polyneuropathy (FAP) Stage [Count of Participants; unit: Participants]
  FAP Stage I: Unimpaired ambulation | 24
  FAP Stage II: Assistance with ambulation required | 3
  FAP Stage III: Wheelchair-bound or bedridden | 0

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Experiencing Adverse Events (AEs), Serious Adverse Events (SAEs) and Study Drug Discontinuation
Description: An AE is any untoward medical occurrence in a patient or clinical investigational patient administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Time Frame: From Baseline up to 56 days post last dose
Population: Safety Analysis Set: All participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | ALN-TTR02 (Patisiran)
Number analyzed (Participants) | 27
participants
  At least 1 Treatment Emergent Adverse Event (TAE) | 26
  At least 1 Serious Adverse Event (SAE) | 7
  Study Drug Discontinuation for any reason | 2

2. Secondary Outcome: Percentage Change From Baseline in Serum TTR Levels
Description: TTR levels, measured using the enzyme-linked immunosorbent assay (ELISA) method.
Time Frame: From Baseline up to 56 days post last dose
Population: Full Analysis Set: All participants who were enrolled were included in the full analysis set.
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | ALN-TTR02 (Patisiran)
Number analyzed (Participants) | 27
Percent Change
  Individual TTR % change | -82.06 (1.33)
  Individual Predose TTR % change | -79.73 (1.45)
  Individual Max TTR % change | -92.54 (0.67)

3. Secondary Outcome: Change From Baseline in the Modified Neuropathy Impairment Score +7 (mNIS+7)
Description: The mNIS+7 assessment is a composite measure of neurologic impairment that provides a comprehensive measure of large and small fiber function that encompasses the totality of the motor, sensory, and autonomic deficits seen in hereditary transthyretin-mediated amyloidosis (hATTR) patients with polyneuropathy. The minimum and maximum values are 0 and 304, respectively. A higher score indicates a worse outcome.
Time Frame: Baseline, Month 24
Population: Full Analysis Set: All participants who were enrolled were included in the full analysis set. The number of participants analyzed is the number for whom evaluable data were available.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | ALN-TTR02 (Patisiran)
Number analyzed (Participants) | 27
score on a scale
  Baseline | 50.5 [2.00 to 122.50]
  Change from Baseline at Month 24: number analyzed (Participants) | 26
  Change from Baseline at Month 24 | -7.00 [-34.63 to 15.38]

4. Secondary Outcome: Change From Baseline in Quality of Life and Disability as Assessed by the EuroQoL (Quality of Life)-5 Dimensions (EQ-5D), EuroQoL Visual Analog Scale (EQ-VAS) Questionnaires and Rasch-built Overall Disability Scale (R-ODS)
Description: The overall EQ-5D is measured on a scale from 0 to 1, with 0 being worst and 1 best. The EQ-VAS is measured on a scale of 0-100, with 0 being the worst and 100 the best. The R-ODS captures activity and social participation limitations in patients. The R-ODS score ranges from 0 (most severe activity and social participation limitations) to 100 (no activity and social participation limitations).
Time Frame: Baseline, Month 24
Population: as for outcome 3
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | ALN-TTR02 (Patisiran)
Number analyzed (Participants) | 27
Score on a scale
  EQ-5D Score at Baseline | 0.76 [0.31 to 1.00]
  EQ-5D Score: Change from Baseline at Month 24: number analyzed (Participants) | 26
  EQ-5D Score: Change from Baseline at Month 24 | 0.00 [-0.22 to 0.17]
  EQ-VAS Score at Baseline | 70.0 [30 to 98]
  EQ-VAS Score: Change from Baseline at Month 24: number analyzed (Participants) | 26
  EQ-VAS Score: Change from Baseline at Month 24 | 0.0 [-25 to 30]
  R-ODS Score at Baseline: number analyzed (Participants) | 26
  R-ODS Score at Baseline | 38.5 [15 to 48]
  R-ODS Score: Change from Baseline at Month 24: number analyzed (Participants) | 25
  R-ODS Score: Change from Baseline at Month 24 | -1.0 [-14 to 8]

5. Secondary Outcome: Change in Gait Speed With 10-meter Walk Test
Description: The 10-meter walk test measures the time (in seconds) that it takes a patient to walk 10 meters.
Time Frame: Baseline, Month 24
Population: as for outcome 3
Measure: Median (Full Range); unit: m/sec
Arm/Group | ALN-TTR02 (Patisiran)
Number analyzed (Participants) | 22
m/sec
  Baseline | 1.13 [0.4 to 2.2]
  Change from Baseline at Month 24: number analyzed (Participants) | 21
  Change from Baseline at Month 24 | 0.09 [-0.4 to 0.3]

6. Secondary Outcome: Mean Change From Baseline in Hand Grip Strength
Description: The mean (SEM) hand grip strength change from baseline at 24 months between patients who used patisiran with or without a concomitant TTR stabilizer.
Time Frame: Baseline, Month 24
Population: as for outcome 3
Measure: Median (Full Range); unit: kg
Arm/Group | ALN-TTR02 (Patisiran)
Number analyzed (Participants) | 27
kg
  Baseline | 23.88 [3.2 to 49.3]
  Change from Baseline at Month 24: number analyzed (Participants) | 26
  Change from Baseline at Month 24 | 1.54 [-17.2 to 22.7]

7. Secondary Outcome: Change From Baseline in Nutritional Status (Modified Body Mass Index, mBMI)
Description: Nutritional status of patients was evaluated using the mBMI, calculated as BMI (kg/m^2) multiplied by albumin (g/L). An increase from baseline in mBMI suggests improvement, and a decrease from baseline suggests worsening.
Time Frame: Baseline, Month 24
Population: as for outcome 3
Measure: Median (Full Range); unit: kg/m^2 x albumin g/L
Arm/Group | ALN-TTR02 (Patisiran)
Number analyzed (Participants) | 27
kg/m^2 x albumin g/L
  Baseline | 1049.09 [728.6 to 1379.6]
  Change from Baseline at Month 24: number analyzed (Participants) | 22
  Change from Baseline at Month 24 | -39.85 [-368.8 to 258.9]

ADVERSE EVENTS:
Time Frame: The investigators reported all AEs that occurred after the start of study drug administration on Day 0 (Baseline) through 21 or 56 days after the last dose of study drug administration (depending on enrollment into the open-label global extension study).
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study
Groups:
- Safety Population: All patients who received at least one dose of ALN-TTR02 (patisiran)
Arm/Group | Safety Population
All-Cause Mortality (participants affected / at risk) | 2/27
Serious Adverse Events (participants affected / at risk) | 7/27
Other Adverse Events (participants affected / at risk) | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=27)
Cardiac amyloidosis (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Abscess limb (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute prerenal failure (Renal and urinary disorders) | 1
Arthrodesis (Surgical and medical procedures) | 1
Venous thrombosis limb (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=27)
Flushing (Vascular disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 6
Infusion related reaction (Immune system disorders) | 6
Nasopharyngitis (Infections and infestations) | 6
Vomiting (Gastrointestinal disorders) | 6
Wound (Injury, poisoning and procedural complications) | 6
Nausea (Gastrointestinal disorders) | 5
Urinary tract infection (Infections and infestations) | 5
Insomnia (Psychiatric disorders) | 4
Neuralgia (Nervous system disorders) | 4
Pyrexia (General disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 3
Bronchitis (Infections and infestations) | 3
Cataract (Eye disorders) | 3
Infusion site extravasation (General disorders) | 3
Macular degeneration (Eye disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Oedema peripheral (General disorders) | 3
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3
Macular fibrosis (Eye disorders) | 2
Visual acuity reduced (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Early satiety (General disorders) | 2
Fatigue (General disorders) | 2
Gait disturbance (General disorders) | 2
Infusion site erythema (General disorders) | 2
Pain (General disorders) | 2
Cellulitis (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 2
Wound infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 2
Foot fracture (Injury, poisoning and procedural complications) | 2
Blood thyroid stimulating hormone decreased (Investigations) | 2
Weight decreased (Investigations) | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 2
Visual field defect (Nervous system disorders) | 2
Depression (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2015-06-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT01961921/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT01961921/SAP_001.pdf